CLINICAL TRIAL: NCT04351061
Title: Pilot Study of Acetazolamide to Prevent Post Operative Cerebrospinal Fluid (CSF) Leak in Patients Undergoing Endoscopic Skull Base Surgery
Brief Title: Acetazolamide for the Prevention of Post Operative CSF Leak
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants were identified per inclusion/exclusion criteria
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ronald Benveniste, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20191265
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Cerebrospinal Fluid Leak
MeSH Terms: conditions — Cerebrospinal Fluid Leak | interventions — Acetazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acetazolamide Arm (Experimental): Participants in this arm will receive the Acetazolamide intervention for 7 consecutive days post standard of care endoscopic skull base surgery.
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide 500 mg by mouth twice per day for 7 consecutive days.
  Other Names: Diamox

SUMMARY:
The purpose of this research is to test the use of Acetazolamide in preventing post-operative cerebrospinal fluid leak in patients having endoscopic skull base surgery (it is a surgery performed through the nose and sinus).

ELIGIBILITY:
Inclusion Criteria:

* Elective transsphenoidal resection of a tumor expected to result in an intraoperative high flow CSF leak; such tumors include craniopharyngioma, meningioma, and Rathke cleft cyst.
* Elective transsphenoidal resection of a pituitary adenoma, with BMI >25, or with observed low or high flow CSF leak during surgery, conferring an elevated risk of postoperative CSF leak.
* Patients who voluntarily sign Informed Consent
* Male subjects and female subjects of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception during study treatment and for at least 1 month after stopping study treatment. Male subjects should refrain from donating semen during treatment and 1 month after stopping treatment.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Patients with prior adverse reactions to acetazolamide or who are taking aspirin concomitantly (which may increase the risk of adverse reactions to acetazolamide)
* Patients with moderate to severe chronic obstructive pulmonary disease (which may increase the risk of adverse effects of acetazolamide)
* Acetazolamide therapy is contraindicated in situations in which sodium and/or potassium blood serum levels are depressed, in cases of marked kidney and liver disease or dysfunction, in suprarenal gland failure, and in hyperchloremic acidosis.
* It is contraindicated in patients with cirrhosis because of the risk of development of hepatic encephalopathy
* Sulfonamide allergy
* Pregnant females, breastfeeding females, and males and females of childbearing potential who are unwilling or unable to use a highly effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Incidence of CSF Leakage | 30 days
  Occurrence of post operative CSF leak within 30 days of surgery confirmed on clinical examination as well on CT scan, endoscopic evaluation or confirmation via beta transferrin testing

SECONDARY OUTCOMES:
Incidence of suspected drug events | 14 days
  Treatment emergent adverse events as assessed by treating physician discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Benveniste, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No